CLINICAL TRIAL: NCT00444080
Title: A Multi Center Study Comparing the Ex-PRESSTM Mini Glaucoma Shunt to Trabeculectomy in Subjects With Open Angle Glaucoma
Brief Title: Comparison of Ex-PRESSTM Mini Glaucoma Shunt to Trabeculectomy in Subjects With Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Peter Netland, MD, Vernah Scott Moyston Professor, Chair, Department of Ophthalmology, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14967
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Glaucoma
Keywords: Ex-PRESS; TRABECULECTOMY
MeSH Terms: conditions — Glaucoma | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (Active Comparator): Subjects undergoing trabeculectomy with the use of Mitomycin C
  Interventions: Procedure: Trabeculectomy
- Treatment Arm (Experimental): Subjects undergoing Ex-PRESS Under Scleral Flap implantation procedure with the use of Mitomycin C
  Interventions: Device: Ex-PRESS mini shunt

INTERVENTIONS:
Procedure: Trabeculectomy — Standard trabeculectomy procedure
  1. Creation of a fornix or limbal based conjunctival flap in upper quadrants
  2. Creation of a limbal-based scleral flap extending into clear cornea
  3. Delicate application of MMC solution onto sclerectomy bed. (MMC concentration 0.4mg/ml for 1-3 minutes)
  4. Creation of fistula 1mm x 2mm in size
  5. Iridectomy
  6. Suturing the scleral flap
  7. Repositioning of conjunctiva with sutures After procedure, antibiotics & steroids are administered topically; eye is covered with a pad - patient is discharged.
  Arms: Control Arm
Device: Ex-PRESS mini shunt — Ex-PRESS implantation procedure:
  1. Creation of a fornix or limbal based conjunctival flap in upper quadrants
  2. Creation of limbal-based scleral flap extending into clear cornea
  3. Delicate application of MMC solution onto sclerectomy bed. (MMC concentration 0.4mg/ml for 1-3 minutes)
  4. Penetration into anterior chamber using 23-25G needle, halfway between the white sclera and clear cornea (in the center of the grey zone);creation of track incision at limbus
  5. Prior to implantation, a thorough mobility check should be performed
  6. Implantation of Ex-PRESS implant loaded on its introducer, through that pre-incision
  7. Withdrawal of introducer
  8. Tucking plate under the scleral flap, and verification of its position
  9. Suturing scleral flap After implantation procedure, antibiotics & steroids administered topically; eye is covered with a pad - patient is discharged.
  Arms: Treatment Arm

SUMMARY:
A prospective randomized trial to compare the safety and efficacy of the Ex-PRESS to trabeculectomy in patients with open angle glaucoma who failed medical or are allergic to medical treatment and for which filtering surgery is indicated. Surgical success was defined as 5 mmHg ≤ intraocular pressure ≤ 18 mmHg, with or without medications, without further glaucoma surgery. Postoperative intraocular pressure, number of medications, complications and success rates were followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject over the age of 18
* Subject diagnosed with open angle glaucoma (POAG, PXFG or PDSG) or ocular hypertension
* Subject is a candidate for filtering surgery with intraoperative anti-metabolites
* IOP > 18 mmHg on maximum tolerated medial therapy based on two measurements taken 1 hour apart at the same visit.
* Subject willing to attend all follow-up evaluations
* Subject willing to sign informed consent.

Exclusion Criteria:

* Subject diagnosed with: PACG, NTG, secondary glaucoma, neovascular glaucoma
* Subject has history of glaucoma surgery (filtering, glaucoma drainage device, cyclo destructive procedures)
* Subject has history of penetrating keratoplasty (PKP)
* Subject underwent large incision extra capsular cataract extraction
* Subject had cataract phacoemulsification within the last month
* Subject has a visually significant cataract that is planned for extraction at the time of filtering surgery or within 12 months thereafter
* Any ocular disease or history in the operated eye other than glaucoma and cataract, such as uveitis, ocular infection, severe dry eye, severe blepharitis , active proliferative retinopathy, ICE syndrome, epithelial or fibrous down growth, aphakia, and ocular pathology that may interfere with accurate IOP measurements
* Subject has vitreous present in the anterior chamber for which vitrectomy is anticipated
* IOP of ≤18mmHg
* Subject participates in any other concurrent ocular investigation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Netland, MD, PhD, Principal Investigator — University of Virginia
Locations (8):
- United States (7):
  - University of California, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Washington University, St Louis, Missouri
  - Dean A. McGee Eye Institute, Oklahoma City, Oklahoma
  - Wills EYE Institute, Philadelphia, Pennsylvania
  - Allegheny Ophthalmic & Orbital Associates, P.C., Pittsburgh, Pennsylvania
  - University of Tennessee, Memphis, Tennessee
- Osler Eyecare, Mississauga, Ontario, Canada

REFERENCES:
- [Result] Netland PA, Sarkisian SR Jr, Moster MR, Ahmed II, Condon G, Salim S, Sherwood MB, Siegfried CJ. Randomized, prospective, comparative trial of EX-PRESS glaucoma filtration device versus trabeculectomy (XVT study). Am J Ophthalmol. 2014 Feb;157(2):433-440.e3. doi: 10.1016/j.ajo.2013.09.014. Epub 2013 Nov 7. PMID 24210765
- [Derived] Park J, Rittiphairoj T, Wang X, E JY, Bicket AK. Device-modified trabeculectomy for glaucoma. Cochrane Database Syst Rev. 2023 Mar 13;3(3):CD010472. doi: 10.1002/14651858.CD010472.pub3. PMID 36912740
- See also: Study results indexed on Pub Med — https://pubmed.ncbi.nlm.nih.gov/24210765/

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: Subjects undergoing trabeculectomy with the use of Mitomycin C
  Trabeculectomy: Standard trabeculectomy procedure
  1. Creation of a fornix or limbal based conjunctival flap in upper quadrants
  2. Creation of a limbal-based scleral flap extending into clear cornea
  3. Delicate application of MMC solution onto sclerectomy bed. (MMC concentration 0.4mg/ml for 1-3 minutes)
  4. Creation of fistula 1mm x 2mm in size
  5. Iridectomy
  6. Suturing the scleral flap
  7. Repositioning of conjunctiva with sutures After procedure, antibiotics & steroids are administered topically; eye is covered with a pad - patient is discharged.
- Treatment Arm: Subjects undergoing Ex-PRESS Under Scleral Flap implantation procedure with the use of Mitomycin C
  Ex-PRESS mini shunt: Ex-PRESS implantation procedure:
  1. Creation of a fornix or limbal based conjunctival flap in upper quadrants
  2. Creation of limbal-based scleral flap extending into clear cornea
  3. Delicate application of MMC solution onto sclerectomy bed. (MMC concentration 0.4mg/ml for 1-3 minutes)
  4. Penetration into anterior chamber using 23-25G needle, halfway between the white sclera and clear cornea (in the center of the grey zone);creation of track incision at limbus
  5. Prior to implantation, a thorough mobility check should be performed
  6. Implantation of Ex-PRESS implant loaded on its introducer, through that pre-incision
  7. Withdrawal of introducer
  8. Tucking plate under the scleral flap, and verification of its position
  9. Suturing scleral flap After implantation procedure, antibiotics & steroids administered topically; eye is covered with a pad.
Period: Overall Study
Arm/Group | Control Arm | Treatment Arm
Started | 61 | 59
Completed | 61 | 59
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Treatment Arm | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 23 | 48
  >=65 years | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (11.6) | 67.8 (10.4) | 68.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 33 | 32 | 65
Region of Enrollment [Number; unit: participants]
  United States | 55 | 52 | 107
  Canada | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Intraocular Pressure
Description: Mean postoperative intraocular pressure
Time Frame: assessed at 1d, 1w, 1m, 3m, 6m, 12m, 18m, 24m. 24 months reported
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Groups:
- Treatment Arm: Subjects undergoing Ex-PRESS Under Scleral Flap implantation procedure with the use of Mitomycin C
  Ex-PRESS mini shunt procedure:
  1. Creation of a fornix or limbal based conjunctival flap in upper quadrants
  2. Creation of limbal-based scleral flap extending into clear cornea
  3. Delicate application of MMC solution onto sclerectomy bed. (MMC concentration 0.4mg/ml for 1-3 minutes)
  4. Penetration into anterior chamber using 23-25G needle, halfway between the white sclera and clear cornea (in the center of the grey zone);creation of track incision at limbus
  5. Prior to implantation, a thorough mobility check should be performed
  6. Implantation of Ex-PRESS implant loaded on its introducer, through that pre-incision
  7. Withdrawal of introducer
  8. Tucking plate under the scleral flap, and verification of its position
  9. Suturing scleral flap After implantation procedure, antibiotics & steroids administered topically; eye is covered with a pad - patient is discharged.
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 61 | 59
Number analyzed (eyes) | 61 | 59
mmHg | 14.6 (7.1) | 14.7 (4.6)

2. Primary Outcome: Medications
Time Frame: assessed at 1d, 1w, 1m, 3m, 6m, 12m, 18m, 24m; 24 months reported
Measure: Mean (Standard Deviation); unit: number of medications
Units Other Than Participants: eyes
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 61 | 59
Number analyzed (eyes) | 61 | 59
number of medications | 0.7 (1.2) | 0.9 (1.3)

3. Secondary Outcome: Safety - Incidence of Adverse Events
Description: Comparison of the incidence of all adverse events that occur during the intra-operative and postoperative periods between the two study arms. More than 1 complication may have occurred in the same subject.
Time Frame: 24 months
Measure: Number; unit: complications
Units Other Than Participants: eyes
Groups:
- Treatment Arm: Subjects undergoing Ex-PRESS Under Scleral Flap implantation procedure with the use of Mitomycin C
  Ex-PRESS mini shunt implantation procedure:
  1. Creation of a fornix or limbal based conjunctival flap in upper quadrants
  2. Creation of limbal-based scleral flap extending into clear cornea
  3. Delicate application of MMC solution onto sclerectomy bed. (MMC concentration 0.4mg/ml for 1-3 minutes)
  4. Penetration into anterior chamber using 23-25G needle, halfway between the white sclera and clear cornea (in the center of the grey zone);creation of track incision at limbus
  5. Prior to implantation, a thorough mobility check should be performed
  6. Implantation of Ex-PRESS implant loaded on its introducer, through that pre-incision
  7. Withdrawal of introducer
  8. Tucking plate under the scleral flap, and verification of its position
  9. Suturing scleral flap After implantation procedure, antibiotics & steroids administered topically; eye is covered with a pad - patient is discharged.
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 61 | 59
Number analyzed (eyes) | 61 | 59
complications | 25 | 11
Statistical Analysis 1: Comparison: Control Arm vs Treatment Arm; Test type: Other; p = 0.013, Fisher Exact

4. Secondary Outcome: Efficacy - The Number of Participants With Qualified and Complete Success
Description: The secondary effectiveness measure will be qualified and complete success rate defined as IOP≤18mmHg with or without medications in the test group as compared to qualified and complete success rate in the concurrent control group at 24 month
Time Frame: 24 months
Measure: Number; unit: participants
Units Other Than Participants: eyes
Arm/Group | Control Arm | Treatment Arm
Number analyzed (Participants) | 61 | 59
Number analyzed (eyes) | 61 | 59
participants | 48 | 49

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Control Arm | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/59
Other Adverse Events (participants affected / at risk) | 22/61 | 9/59
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=61) | Treatment Arm (N=59)
Shallow anterior chamber (Eye disorders) | 7 (7) | 4 (4)
Surgically treated cataract (Eye disorders) | 7 (7) | 3 (3)
Hyphema (Eye disorders) | 6 (6) | 0 (0)
Early wound leak (Eye disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-09-05): https://cdn.clinicaltrials.gov/large-docs/80/NCT00444080/Prot_SAP_000.pdf